CLINICAL TRIAL: NCT00409617
Title: A Multi-Center, Open-Label Study of the Fully Human Anti-TNF Monoclonal Antibody Adalimumab for the Induction and Maintenance of Clinical Remission in Subjects With Moderate to Severe Crohn's Disease
Brief Title: Study of Adalimumab Treatment for Induction and Maintenance of Clinical Remission in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-829; EudraCT:2006-002078-23
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Adalimumab 40 mg Every Other Week dosing
  Other Names: Humira
Biological: adalimumab — Adalimumab 40 mg Every Week dosing if participant experiences a disease flare or is not responding to treatment. A disease flare is defined as an increase of 3 points or more on the HBI compared to the Baseline score and a total HBI score of 7 or higher. Non-response is defined as a decrease by fewer than 3 points in the HBI compared to Baseline.
  Other Names: Humira

SUMMARY:
The purpose of this study is to evaluate the safety of adalimumab for treatment of patients with moderate to severe Crohn's Disease (CD) and to measure the effects of treatment on patient general well-being, health-related quality of life (QoL), fistula healing, CD-related extra-intestinal manifestations, work performance, and overall activity.

DETAILED DESCRIPTION:
This is an open-label, multi-center, study designed to evaluate the safety and efficacy of adalimumab on inducing and maintaining clinical remission in subjects with moderate to severe Crohn's Disease.

Approximately 1000 subjects with a diagnosis of moderate to severe Crohn's Disease (Harvey Bradshaw Index score >= 7) will be enrolled at approximately 200 sites within Europe. Enrollment will be dependent on meeting all screening criteria.

Study medication will be administered by subcutaneous injection. At Baseline (Week 0), all subjects will receive a dose of 160 mg adalimumab. At Week 2, all subjects will receive a dose of 80 mg adalimumab. Starting at Week 4, all subjects will begin receiving injections of adalimumab 40 mg every other week and will continue every other week dosing through Week 20 except in the case of disease flare or non-response.

Starting at Week 12, subjects who experience a disease flare (flare is defined by an increase in the Harvey Bradshaw Index >=3 and a total Index score of >=7 when compared to Week 4) or are not responding to adalimumab treatment (non-response is defined as a decrease in the Harvey Bradshaw Index by fewer than 3 points compared to Baseline) will be permitted to increase study therapy to adalimumab 40 mg every week.

If the subject continues to demonstrate a lack of improvement on every week adalimumab therapy, they may be withdrawn from the study.

Prior to Week 8 subjects will not be allowed to increase or decrease Crohn's specific concomitant medications except in the event of concomitant Crohn's treatment-related toxicities assessed as moderate to severe. Changes in concomitant medications at/after Week 8 will be at the Investigator's discretion.

Subjects will be evaluated for safety and efficacy at Baseline (Week 0), Weeks 2, 4, 8, 12, and 20, and at unscheduled visits. Efficacy evaluations include HBI, Short Inflammatory Bowel Disease Questionnaire (SIBDQ), Work Productivity Activity Index (WPAI) questionnaire, fistula counts, health care resource utilization (HCRU), and evaluation of CD-related extra-intestinal manifestations (EIMs). Safety assessments include vital signs, physical examination, general laboratory analyses, urinalysis, and monitoring of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe Crohn's Disease confirmed by endoscopy or radiologic evaluation for greater than 4 months (16 weeks)
* Inadequate response to conventional therapy for Crohn's Disease
* Subjects >=18 and <=75 years of age and in good health (Investigator discretion) with a recent stable medical history
* Harvey Bradshaw Index score of 7 or higher

Exclusion Criteria:

* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Subject who has had surgical bowel resections within the past 6 months or is planning any resection at any time point while enrolled in the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant
* Previous treatment with adalimumab or previous participation in an adalimumab clinical study
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Subjects with any prior exposure to Tysabri® (natalizumab)
* Subjects on prednisone >40 mg/day (or equivalent), subjects on budesonide >9 mg/day, or subjects who are taking prednisone and budesonide concurrently at Baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pollack, MD, Study Director — Abbott
Locations (189):
- Austria (5):
  - Site Ref # / Investigator 3077, Graz
  - Site Ref # / Investigator 2978, Vienna
  - Site Ref # / Investigator 2975, Vienna
  - Site Ref # / Investigator 2976, Vienna
  - Site Ref # / Investigator 2977, Wels
- Belgium (8):
  - Site Ref # / Investigator 3023, Bonheiden
  - Site Ref # / Investigator 3021, Brussels
  - Site Ref # / Investigator 3074, Brussels
  - Site Ref # / Investigator 3020, Edegem
  - Site Ref # / Investigator 3625, Ghent
  - Site Ref # / Investigator 3773, Leuven
  - Site Ref # / Investigator 3022, Liège
  - Site Ref # / Investigator 3047, Roeselare
- Czechia (4):
  - Site Ref # / Investigator 3893, Brno
  - Site Ref # / Investigator 4657, Olomouc
  - Site Ref # / Investigator 4660, Prague
  - Site Ref # / Investigator 4659, Prague
- Denmark (5):
  - Site Ref # / Investigator 3075, Aalborg
  - Site Ref # / Investigator 3037, Aarhus C
  - Site Ref # / Investigator 3088, Elsinore
  - Site Ref # / Investigator 3076, Hvidovre
  - Site Ref # / Investigator 3019, Odense C
- Site Ref # / Investigator 3623, Hyvinkää, Finland
- France (30):
  - Site Ref # / Investigator 3032, Amiens
  - Site Ref # / Investigator 3012, Besançon
  - Site Ref # / Investigator 2983, Béthune
  - Site Ref # / Investigator 2993, Bordeaux
  - Site Ref # / Investigator 2982, Caen
  - Site Ref # / Investigator 3015, Clichy
  - Site Ref # / Investigator 3011, Colombes
  - Site Ref # / Investigator 3030, Créteil
  - Site Ref # / Investigator 3033, Créteil
  - Site Ref # / Investigator 3027, Évry
  - Site Ref # / Investigator 3048, Grenoble
  - Site Ref # / Investigator 3097, Lille
  - Site Ref # / Investigator 3031, Marseille
  - Site Ref # / Investigator 2985, Montfermeil
  - Site Ref # / Investigator 2994, Montpellier
  - Site Ref # / Investigator 3014, Nantes
  - Site Ref # / Investigator 3029, Nice
  - Site Ref # / Investigator 3017, Paris
  - Site Ref # / Investigator 2995, Paris
  - Site Ref # / Investigator 3025, Paris
  - Site Ref # / Investigator 2996, Paris
  - Site Ref # / Investigator 3016, Paris
  - Site Ref # / Investigator 4275, Paris
  - Site Ref # / Investigator 3026, Pessac
  - Site Ref # / Investigator 2974, Pierre-Bénite
  - Site Ref # / Investigator 3013, Reims
  - Site Ref # / Investigator 3024, Rouen
  - Site Ref # / Investigator 2973, Strasbourg
  - Site Ref # / Investigator 2986, Toulouse
  - Site Ref # / Investigator 3018, Vandœuvre-lès-Nancy
- Germany (48):
  - Site Ref # / Investigator 2969, Augsburg
  - Site Ref # / Investigator 3096, Berlin
  - Site Ref # / Investigator 3041, Berlin
  - Site Ref # / Investigator 3070, Berlin
  - Site Ref # / Investigator 2980, Berlin
  - Site Ref # / Investigator 3089, Berlin
  - Site Ref # / Investigator 3084, Bochum
  - Site Ref # / Investigator 3051, Bochum
  - Site Ref # / Investigator 3086, Braunschweig
  - Site Ref # / Investigator 3094, Cottbus
  - Site Ref # / Investigator 2972, Dachau
  - Site Ref # / Investigator 3053, Dresden
  - Site Ref # / Investigator 3368, Düren
  - Site Ref # / Investigator 3052, Erlangen
  - Site Ref # / Investigator 3085, Essen
  - Site Ref # / Investigator 3092, Frankfurt
  - Site Ref # / Investigator 3040, Freiburg im Breisgau
  - Site Ref # / Investigator 3066, Halle
  - Site Ref # / Investigator 2981, Hamburg
  - Site Ref # / Investigator 3044, Hamburg
  - Site Ref # / Investigator 2979, Hamburg
  - Site Ref # / Investigator 3043, Hamburg
  - Site Ref # / Investigator 3082, Hamburg
  - Site Ref # / Investigator 3081, Hanover
  - Site Ref # / Investigator 3072, Heidelberg
  - Site Ref # / Investigator 3093, Herne
  - Site Ref # / Investigator 3080, Jena
  - Site Ref # / Investigator 3034, Karlsruhe
  - Site Ref # / Investigator 3617, Kiel
  - Site Ref # / Investigator 3071, Leipzig
  - Site Ref # / Investigator 3091, Lübeck
  - Site Ref # / Investigator 3090, Magdeburg
  - Site Ref # / Investigator 3049, Mainz
  - Site Ref # / Investigator 3083, Mainz
  - Site Ref # / Investigator 3073, Mannheim
  - Site Ref # / Investigator 3050, Minden
  - Site Ref # / Investigator 3098, Munich
  - Site Ref # / Investigator 3055, Munich
  - Site Ref # / Investigator 3054, Munich
  - Site Ref # / Investigator 3056, Münster
  - Site Ref # / Investigator 3057, Münster
  - Site Ref # / Investigator 3046, Osnabrück
  - Site Ref # / Investigator 3078, Regensburg
  - Site Ref # / Investigator 3095, Rostock
  - Site Ref # / Investigator 2970, Rottenburg
  - Site Ref # / Investigator 3042, Stade
  - Site Ref # / Investigator 3045, Stuttgart
  - Site Ref # / Investigator 3079, Stuttgart
- Greece (8):
  - Site Ref # / Investigator 4352, Athens
  - Site Ref # / Investigator 4357, Athens
  - Site Ref # / Investigator 4358, Athens
  - Site Ref # / Investigator 4606, Heraklion
  - Site Ref # / Investigator 4355, Ioannina
  - Site Ref # / Investigator 4353, Nikaia
  - Site Ref # / Investigator 4359, Thessaloniki
  - Site Ref # / Investigator 4351, Thessaloniki
- Ireland (3):
  - Site Ref # / Investigator 3326, Cork
  - Site Ref # / Investigator 3324, Dublin
  - Site Ref # / Investigator 3325, Dublin
- Italy (13):
  - Site Ref # / Investigator 3953, Bologna
  - Site Ref # / Investigator 3061, Florence
  - Site Ref # / Investigator 3035, Milan
  - Site Ref # / Investigator 3065, Naples
  - Site Ref # / Investigator 3036, Padua
  - Site Ref # / Investigator 3062, Palermo
  - Site Ref # / Investigator 3063, Pavia
  - Site Ref # / Investigator 3058, Pescara
  - Site Ref # / Investigator 3064, Rome
  - Site Ref # / Investigator 2991, Rome
  - Site Ref # / Investigator 3039, Rome
  - Site Ref # / Investigator 3087, Rozzano
  - Site Ref # / Investigator 3038, San Donato Milanese
- Norway (5):
  - Site Ref # / Investigator 3618, Bergen
  - Site Ref # / Investigator 3629, Bodø
  - Site Ref # / Investigator 3630, Hamar
  - Site Ref # / Investigator 3620, Oslo
  - Site Ref # / Investigator 3619, Oslo
- Portugal (4):
  - Site Ref # / Investigator 3596, Braga
  - Site Ref # / Investigator 3069, Coimbra
  - Site Ref # / Investigator 4972, Lisbon
  - Site Ref # / Investigator 3068, Lisbon
- Slovakia (3):
  - Site Ref # / Investigator 3493, Bratislava
  - Site Ref # / Investigator 4626, Košice
  - Site Ref # / Investigator 3494, Prešov
- Spain (20):
  - Site Ref # / Investigator 3448, Alicante
  - Site Ref # / Investigator 3009, Badalona - Barcelona
  - Site Ref # / Investigator 3005, Barakaldo
  - Site Ref # / Investigator 2990, Barcelona
  - Site Ref # / Investigator 2989, Barcelona
  - Site Ref # / Investigator 3002, Barcelona
  - Site Ref # / Investigator 3486, Barcelona
  - Site Ref # / Investigator 2998, Cabuenes-Gijon
  - Site Ref # / Investigator 2988, Galdakano
  - Site Ref # / Investigator 4383, Las Palmas de Gran Canaria
  - Site Ref # / Investigator 3484, Madrid
  - Site Ref # / Investigator 2997, Madrid
  - Site Ref # / Investigator 2999, Madrid
  - Site Ref # / Investigator 3447, Madrid
  - Site Ref # / Investigator 3595, Madrid
  - Site Ref # / Investigator 3008, Palma de Mallorca
  - Site Ref # / Investigator 3000, Santander
  - Site Ref # / Investigator 3003, Valencia
  - Site Ref # / Investigator 3007, Zaragoza
  - Site Ref # / Investigator 3010, Zaragoza
- Sweden (10):
  - Site Ref # / Investigator 3895, Gothenburg
  - Site Ref # / Investigator 3500, Gothenburg
  - Site Ref # / Investigator 3499, Linköping
  - Site Ref # / Investigator 3488, Lund
  - Site Ref # / Investigator 3892, Östersund
  - Site Ref # / Investigator 3498, Skövde
  - Site Ref # / Investigator 3489, Stockholm
  - Site Ref # / Investigator 3896, Stockholm
  - Site Ref # / Investigator 3487, Stockholm
  - Site Ref # / Investigator 3594, Umeå
- Switzerland (4):
  - Site Ref # / Investigator 3323, Basel
  - Site Ref # / Investigator 3321, Bern
  - Site Ref # / Investigator 3322, Lausanne
  - Site Ref # / Investigator 3794, Zurich
- United Kingdom (18):
  - Site Ref # / Investigator 4604, Barnstaple
  - Site Ref # / Investigator 4590, Cardiff
  - Site Ref # / Investigator 4603, Dundee
  - Site Ref # / Investigator 4579, Edinburgh
  - Site Ref # / Investigator 4588, Harrow
  - Site Ref # / Investigator 4586, Liverpool
  - Site Ref # / Investigator 4595, London
  - Site Ref # / Investigator 4607, London
  - Site Ref # / Investigator 4596, London
  - Site Ref # / Investigator 4580, London
  - Site Ref # / Investigator 4591, Nottingham
  - Site Ref # / Investigator 4589, Plymouth
  - Site Ref # / Investigator 4592, Portsmouth
  - Site Ref # / Investigator 4597, Rotherham
  - Site Ref # / Investigator 4584, Sheffield
  - Site Ref # / Investigator 4578, Southampton
  - Site Ref # / Investigator 4598, Stockport
  - Site Ref # / Investigator 4581, Surrey

REFERENCES:
- [Derived] Louis E, Lofberg R, Reinisch W, Camez A, Yang M, Pollack PF, Chen N, Chao J, Mulani PM. Adalimumab improves patient-reported outcomes and reduces indirect costs in patients with moderate to severe Crohn's disease: results from the CARE trial. J Crohns Colitis. 2013 Feb;7(1):34-43. doi: 10.1016/j.crohns.2012.02.017. Epub 2012 Apr 4. PMID 22480772

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Adalimumab 40 mg Every Other Week or Every Week: Participants received adalimumab 160 mg by subcutaneous injection at Week 0 and adalimumab 80 mg by subcutaneous injection at Week 2. Beginning at Week 4 of the study, participants received adalimumab 40 mg every other week. Beginning at Week 12, participants who experienced a disease flare (increase in Harvey Bradshaw Index of 3 or more compared to Week 4 and a total Index score of 7 or higher) and participants who did not respond to every other week treatment (non-response defined as a decrease in HBI by fewer than 3 points compared to Baseline) could switch to adalimumab 40 mg every week.
Period: Overall Study
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Started | 945
Completed | 785
Not Completed | 160
Not completed — Adverse Event | 57
Not completed — Lack of Efficacy | 54
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 24
Not completed — Withdrawal by Subject | 8
Not completed — Administrative reasons | 1
Not completed — Not described | 14

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 945
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 919
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 35.3 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 568
  Male | 377
Region of Enrollment [Number; unit: participants]
  Portugal | 19
  Slovakia (Slovak Republic) | 18
  Greece | 25
  Finland | 5
  Spain | 47
  Ireland | 11
  Austria | 47
  United Kingdom | 73
  Switzerland | 15
  Italy | 64
  France | 141
  Czech Republic | 37
  Belgium | 72
  Denmark | 43
  Germany | 266
  Norway | 27
  Sweden | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Clinical Remission at Treatment Week 20. Clinical Remission Defined as Harvey Bradshaw Index (HBI) Score Less Than 5.
Description: 5-items that assess general well-being, abdominal pain, diarrhea, abdominal mass, and complications. Score is total of 1) subject well-being (0=very well; 4=terrible); 2) abdominal pain (0=none; 3=severe); 3) diarrhea (number of time per day); 4) abdominal mass (0=none; 3=definite and tender); 5) complications (number). Maximum total score for HBI is not specified, is dependent on number of diarrhea times each day and number of complications. Clinical remission = HBI less than 5. Highest total score at Baseline was 47. Missing data were imputed using non-responder imputation (NRI).
Time Frame: Week 20 of treatment
Population: Intent-to-treat (ITT) population, defined as all participants who received at least 1 injection of adalimumab. Missing data were imputed using non-responder imputation; participants who discontinued the study prior to Week 20 and participants with no score on the Harvey-Bradshaw Index (missing value) at Week 20 were counted as "no" for remission.
Measure: Number; unit: Participants
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 945
Participants | 492 (4.26)

2. Secondary Outcome: Number of Participants Who Were Responders at Week 20 of Treatment. A Responder Was Defined as a Participant Who Had a Decrease of 3 or More on the HBI.
Description: 5-items that assess general well-being, abdominal pain, diarrhea, abdominal mass, and complications. Score is total of 1) subject well-being (0=very well; 4=terrible); 2) abdominal pain (0=none; 3=severe); 3) diarrhea (number of time per day); 4) abdominal mass (0=none; 3=definite and tender); 5) complications (number). Participants who had a decrease from Baseline of at least 3 points in HBI total score were considered responders. Missing data were imputed using non-responder imputation (NRI).
Time Frame: Week 20 of treatment
Population: ITT Population, defined as all participants who received at least 1 injection of adalimumab. Missing data were imputed using non-responder imputation; participants who discontinued the study prior to Week 20 and participants with no score on the Harvey-Bradshaw Index (missing value) at Week 20 were counted as "no" for response.
Measure: Number; unit: Participants
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 945
Participants | 658

3. Secondary Outcome: Number of Participants Who Had a Reduction in Number of Draining Fistulas of at Least 50% From Baseline to Week 20
Description: A count of the number of cutaneous fistulas draining was performed during each physical examination. Among participants who had draining fistulas at Baseline, the number of participants who had a reduction in the number of draining fistulas of at least 50% from Baseline to Week 20 of treatment was determined. Fistulas were classified as abdominal or perianal.
Time Frame: Week 20 of treatment
Population: 171 participants in the ITT population (participants who received at least 1 injection of adalimumab) had draining fistulas at baseline. Data were available for 148 of the 171 participants at Week 20 of treatment. Missing values were not imputed.
Measure: Number; unit: Participants
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 148
Participants | 53

4. Secondary Outcome: Number of Participants Who Had Extra-intestinal Manifestations (EIM) at Baseline and Resolution by Week 20.
Description: Number of participants who had EIM at baseline and had resolution of those manifestations at Week 20. EIM were skin lesions, eye lesions, joint complaints, CD-related hepatic disease, thrombosis, and nephrolithiasis. EIMs were determined by physical examination.
Time Frame: Week 20 of treatment
Population: 497 participants who received at least 1 injection of adalimumab (ITT population) had baseline EIM data. Missing data were imputed using non-responder imputation; participants who discontinued the study before Week 20 and participants with missing value at Week 20 were counted as "no" for resolution.
Measure: Number; unit: Participants
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 497
Participants | 346

5. Secondary Outcome: Mean Change in Total Score of Short Inflammatory Bowel Disease Questionnaire (SIBDQ) From Baseline to Week 20
Description: 10-item assessment of health-related quality of life (QoL) in patients with inflammatory bowel disease. Participant marks an option from 1 to 7 for each item. For some items, 1=None of the time; for other items, 1=All of the time. Value for all items are summed. Total score=10 to 70; a high score=good quality of life (QoL). An increase in score indicates improvement. An absolute change in the SIBDQ score of 9 is considered a minimum clinically important difference (MCID) for a patient.
Time Frame: Week 20 of treatment
Population: The ITT population, defined as participants who received at least 1 injection of adalimumab, was used in the analysis. 907 participants had data available for calculating change in total score of SIBDQ. Missing values were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: Change in total score
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 907
Change in total score | 13.2 (13.39)

6. Secondary Outcome: Mean Change in Percent Work Time Missed Due to Crohn's Disease From Baseline to Week 20 of Treatment
Description: Percent Work Time Missed (Absenteeism) due to CD is one component of the Work Productivity and Activity Impairment (WPAI) Questionnaire. Score of 0% = no impairment. A decrease in the mean indicates improvement.
Time Frame: Week 20 of treatment
Population: The ITT population, defined as participants who received at least 1 injection of adalimumab, was used in the analysis. 369 participants had data available for calculating change in Percent Work Time Missed. Missing values were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: Percent of work time missed
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 369
Percent of work time missed | -10.8 (33.47)

7. Secondary Outcome: Mean Change in Percent Impairment While Working From Baseline to Week 20 of Treatment
Description: Percent impairment while working is a component of the Work Productivity and Activity Impairment measure. A score of 0% = no impairment. A decrease in mean score indicates lessening of impairment.
Time Frame: Week 20 of treatment
Population: The ITT population, defined as participants who received at least 1 injection of adalimumab, was used in the analysis. Data were available for 382 participants for the calculation of mean change in Percent Impairment While Working from Baseline to Week 20. Data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: Percent impairment at work
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 382
Percent impairment at work | -20.0 (30.89)

8. Secondary Outcome: Mean Change in Overall Work Productivity and Activity Impairment Score From Baseline to Week 20
Description: 6-items that assess impairment in work productivity and daily activity during the 7 days before the assessment. It measures the percentage of overall impairment in work productivity and daily activity due to CD. A WPAI score of 0% = no impairment and a score of 100% = total loss of work productivity or activity. An absolute change in WPAI score of 7% is considered the minimum clinically important difference (MCID).
Time Frame: Week 20 of treatment
Population: The ITT population, defined as participants who received at least 1 injection of adalimumab, was used in the analysis. Data were available for 346 participants for the calculation of mean change in Overall Impairment from Baseline to Week 20. Data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: Percent total impairment
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 346
Percent total impairment | -21.8 (34.29)

9. Secondary Outcome: Mean Change in Activity Impairment Score From Baseline to Week 20
Description: Daily activity is one component of the Work Productivity and Activity Impairment Questionnaire. 0% = no impairment. A decrease in the mean indicates improvement.
Time Frame: Week 20 of treatment
Population: The ITT population, defined as participants who received at least 1 injection of adalimumab, was used. Data for 902 participants were available for calculating change from Baseline at Week 20 of treatment. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Number analyzed (Participants) | 902
Percent activity impairment | -23.6 (30.58)

ADVERSE EVENTS:
Arm/Group | Open Label Adalimumab 40 mg Every Other Week or Every Week
Serious Adverse Events (participants affected / at risk) | 181
Other Adverse Events (participants affected / at risk) | 395
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Open Label Adalimumab 40 mg Every Other Week or Every Week
CD (Gastrointestinal disorders) | 54/945
Abdominal pain (Gastrointestinal disorders) | 8/945
Perianal abscess (Infections and infestations) | 6/945
Intestinal obstruction (Gastrointestinal disorders) | 5/945
Subileus (Gastrointestinal disorders) | 5/945
Vomiting (Gastrointestinal disorders) | 4/945
Abdominal abscess (Infections and infestations) | 3/945
Anastomotic stenosis (Injury, poisoning and procedural complications) | 3/945
Chest pain (General disorders) | 3/945
Depression (Psychiatric disorders) | 3/945
Dizziness (Nervous system disorders) | 3/945
Fistula discharge (Musculoskeletal and connective tissue disorders) | 3/945
Herpes zoster (Infections and infestations) | 3/945
Hypokalemia (Metabolism and nutrition disorders) | 3/945
Ileal stenosis (Gastrointestinal disorders) | 3/945
Pyrexia (General disorders) | 3/945
Anaemia (Blood and lymphatic system disorders) | 2/945
Leukopenia (Blood and lymphatic system disorders) | 1/945
Lymph node pain (Blood and lymphatic system disorders) | 1/945
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1/945
Angina pectoris (Cardiac disorders) | 1/945
Atrial fibrillation (Cardiac disorders) | 1/945
Cardiovascular disorder (Cardiac disorders) | 1/945
Acute vestibular syndrome (Ear and labyrinth disorders) | 1/945
Anal fistula (Gastrointestinal disorders) | 1/945
Anal skin tags (Gastrointestinal disorders) | 1/945
Colonic stenosis (Gastrointestinal disorders) | 2/945
Diarrhoea (Gastrointestinal disorders) | 1/945
Enteritis (Gastrointestinal disorders) | 1/945
Enterocolonic fistula (Gastrointestinal disorders) | 1/945
Frequent bowel movements (Gastrointestinal disorders) | 1/945
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1/945
Gastrointestinal fistula (Gastrointestinal disorders) | 1/945
Haemorrhoidal haemorrrhage (Gastrointestinal disorders) | 1/945
Ileitis (Gastrointestinal disorders) | 1/945
Ileorectal fistula (Gastrointestinal disorders) | 1/945
Inflammatory bowel disease (Gastrointestinal disorders) | 1/945
Intestinal fistula (Gastrointestinal disorders) | 1/945
Intestinal functional disorder (Gastrointestinal disorders) | 1/945
Intestinal stenosis (Gastrointestinal disorders) | 2/945
Large intestinal ulcer (Gastrointestinal disorders) | 1/945
Nausea (Gastrointestinal disorders) | 2/945
Pancreatitis (Gastrointestinal disorders) | 1/945
Peritonitis (Gastrointestinal disorders) | 1/945
Rectal haemorrhage (Gastrointestinal disorders) | 1/945
Small intestinal obstruction (Gastrointestinal disorders) | 2/945
Small intestinal perforation (Gastrointestinal disorders) | 2/945
Asthenia (Gastrointestinal disorders) | 1/945
Disease progression (General disorders) | 1/945
Influenza like illness (General disorders) | 1/945
Malaise (General disorders) | 1/945
Biliary colic (Hepatobiliary disorders) | 1/945
Cholelithiasis (Hepatobiliary disorders) | 1/945
Hepatomegaly (Hepatobiliary disorders) | 1/945
Portal vein thrombosis (Hepatobiliary disorders) | 1/945
Abdominal wall abscess (Infections and infestations) | 1/945
Abscess (Infections and infestations) | 2/945
Abscess intestinal (Infections and infestations) | 1/945
Anogenital warts (Infections and infestations) | 1/945
Bacterial infection (Infections and infestations) | 1/945
Bronchiectasis (Infections and infestations) | 1/945
Bronchitis (Infections and infestations) | 1/945
Bronchopneumonia (Infections and infestations) | 1/945
Campylobacter intestinal infection (Infections and infestations) | 1/945
Clostridial infection (Infections and infestations) | 2/945
Clostridium difficile colitis (Infections and infestations) | 1/945
Diverticulitis (Infections and infestations) | 2/945
Enteritis infectious (Infections and infestations) | 1/945
Enterocolitis bacterial (Infections and infestations) | 1/945
Epstein-Barr virus infection (Infections and infestations) | 1/945
Folliculitis (Infections and infestations) | 1/945
Gastroenteritis (Infections and infestations) | 2/945
Gastroenteritis viral (Infections and infestations) | 2/945
Infection (Infections and infestations) | 1/945
Klebsiella sepsis (Infections and infestations) | 1/945
Oesophageal candidiasis (Infections and infestations) | 1/945
Pelvic abscess (Infections and infestations) | 1/945
Perineal abscess (Infections and infestations) | 1/945
Perirectal abscess (Infections and infestations) | 1/945
Pharyngitis (Infections and infestations) | 1/945
Pneumonia (Infections and infestations) | 1/945
Pseudomembranous colitis (Infections and infestations) | 1/945
Pyelonephritis (Infections and infestations) | 1/945
Rectal abscess (Infections and infestations) | 2/945
Sepsis (Infections and infestations) | 1/945
Urinary tract infection (Infections and infestations) | 1/945
Viral infection (Infections and infestations) | 1/945
Jaw fracture (Injury, poisoning and procedural complications) | 1/945
Post procedural complication (Injury, poisoning and procedural complications) | 1/945
Rib fracture (Injury, poisoning and procedural complications) | 1/945
Colonoscopy (Investigations) | 1/945
Diagnostic procedure (Investigations) | 1/945
Platelet count decreased (Investigations) | 1/945
Tuberculin test positive (Investigations) | 1/945
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1/945
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/945
Arthritis (Musculoskeletal and connective tissue disorders) | 2/945
Bursitis (Musculoskeletal and connective tissue disorders) | 1/945
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1/945
Fistula (Musculoskeletal and connective tissue disorders) | 2/945
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/945
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/945
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/945
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/945
Myalgia (Musculoskeletal and connective tissue disorders) | 1/945
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1/945
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1/945
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/945
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/945
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/945
Benign intracranial hypertension (Nervous system disorders) | 1/945
Demyelination (Nervous system disorders) | 1/945
Headache (Nervous system disorders) | 2/945
Hypoaesthesia (Nervous system disorders) | 1/945
Lethargy (Nervous system disorders) | 1/945
Neuralgic amyotrophy (Nervous system disorders) | 1/945
Neuropathy peripheral (Nervous system disorders) | 1/945
Syncope (Nervous system disorders) | 1/945
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/568
Panic attack (Psychiatric disorders) | 1/945
Suicide attempt (Psychiatric disorders) | 1/945
Cystitis noninfective (Renal and urinary disorders) | 1/945
Nephritis (Renal and urinary disorders) | 1/945
Nephrolithiasis (Renal and urinary disorders) | 2/945
Renal colic (Renal and urinary disorders) | 1/945
Cervical dysplasia (Reproductive system and breast disorders) | 1/568
Female genital tract fistula (Reproductive system and breast disorders) | 1/568
Menorrhagia (Reproductive system and breast disorders) | 1/568
Metrorrhagia (Reproductive system and breast disorders) | 1/568
Ovarian hemorrhage (Reproductive system and breast disorders) | 1/568
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/945
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/945
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1/945
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1/945
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/945
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/945
Cold sweat (Skin and subcutaneous tissue disorders) | 1/945
Eczema (Skin and subcutaneous tissue disorders) | 2/945
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1/945
Thrombosis (Vascular disorders) | 1/945
Abortion induced (Surgical and medical procedures) | 2/568
Intestinal anastomosis (Surgical and medical procedures) | 1/945
Medical device removal (Surgical and medical procedures) | 1/945
Adrenal insufficiency (Endocrine disorders) | 1/945
Anal abscess (Infections and infestations) | 2/945
Influenza (Infections and infestations) | 1/945
Vaginal infection (Infections and infestations) | 1/568
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Open Label Adalimumab 40 mg Every Other Week or Every Week
Abdominal pain (Gastrointestinal disorders) | 62/945
Crohn's disease (Gastrointestinal disorders) | 56/945
Nausea (Gastrointestinal disorders) | 72/945
Nasopharyngitis (Infections and infestations) | 136/945
Arthralgia (Musculoskeletal and connective tissue disorders) | 72/945
Headache (Nervous system disorders) | 179/945

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide ABBOTT at least thirty (30) days prior to submission for review, ABBOTT shall return comments promptly. Proposed draft shall be delayed an additional sixty (60) days in addition to the Review Period.